CLINICAL TRIAL: NCT00895063
Title: Effect of Vocal Exercise After Botulinum Toxin Injection for Spasmodic Dysphonia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BOTOXEX
Record Dates: First submitted 2009-05-06; First posted 2009-05-07 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Spasmodic Dysphonia; Dystonia
Keywords: Spasmodic Dysphonia; Botulinum Toxin; Vocal Exercise
MeSH Terms: conditions — Dysphonia; Dystonia | interventions — Botulinum Toxins; Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vocal Exercise (Experimental): Subject will speak continually for one hour following injection of botulinum toxin.
  Interventions: Behavioral: Vocal Exercise
- Silence (Placebo Comparator): Subject will remain silent for one hour following injection of botulinum toxin.
  Interventions: Behavioral: Vocal Exercise

INTERVENTIONS:
Behavioral: Vocal Exercise — This project will examine whether or not exercise performed immediately following botulinum toxin injection affects the clinical benefit received from the injection. This is a cross-over study and subjects will be randomly assigned to a group where they will speak continually for one hour or remain silent for one hour following injection. Data on the effectiveness of the exercise will be collected just before each injection and at 2 weeks, 6 weeks, and 3 months following injection.
  Other Names: Botulinum toxin; BOTOX; BTX; BoNT

SUMMARY:
Studies have suggested that voluntary muscle exercise in the hand and face after botulinum toxin injection may enhance the clinical effects of the toxin. Exercise may speed up the absorption of the toxin by the nerves and enhance the clinical response. This study will explore the effect of exercise on botulinum toxin injections for spasmodic dysphonia (SD).

DETAILED DESCRIPTION:
SD is a rare voice disorder that usually starts when individuals are in early adulthood and occurs in two common forms: adductor and abductor (Aronson, 1968, Brin et al., 1992, Schweinfurth et al., 2002). Adductor is the more common form (Aronson, 1985, Blitzer et al. 1998). With adductor SD, patients have been described as "trying to talk whilst being choked" (Critchley, 1939). The spasmodic hyperadduction of the vocal folds is associated with strained-strangled, rough voice quality and sudden intermittent voice arrests (Aminoff, Dedo, & Izdebski, 1978, Blitzer & Brin, 1992, Hillel, 2001, Izdebski 1992, Ludlow, Nauton, & Bassich, 1984, Woodson, Zwirner, Murry, & Swenson, 1991). On the other hand, the intermittent or continuous abduction of the vocal folds linked with abductor SD results in breathy or whispered voice quality with sudden intermittent voice arrests (Aronson, 1985, Hillel, 2001, and Zwitman, 1979).

Local injection of botulinum toxin is an effective treatment for spasmodic dysphonia and The National Academies of Otolaryngology and Neurology has endorsed the toxin as the treatment of choice for adductor spasmodic dysphonia. Consequently, this treatment is widely used. The clinical benefit of the botulinum toxin is related to muscle weakness in the vocal folds and the benefit lasts from 6 weeks to 6 months.

Studies have suggested that voluntary muscle exercise in the hand and face after botulinum toxin injection may enhance the clinical effects of the toxin (Chen, Scott, & Smith, 2002; Chen et al., 1999; Kim et. al 2003;. Exercise may speed up the absorption of the toxin by the nerves and enhance the clinical response. You are invited to take part in a research study to learn more about the effect of exercise on botulinum toxin injections for spasmodic dysphonic. This project will examine whether or not exercise performed immediately following botulinum toxin injection affects the clinical benefit received from the injection.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of adductor spasmodic dysphonia
2. receiving ongoing botulinum toxin injections for a minimum of 1 year
3. improvement in voice to at least 70% following each of the last three injections

Exclusion Criteria:

1. other neurological disorder
2. other dystonia
3. upper respiratory infection in the last two weeks
4. analgesia at time of injection
5. illiterate
6. under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Self-rating of vocal function | Baseline, 2 weeks, 6 weeks, 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Celia F Stewart, Ph.D., Principal Investigator — New York University
Locations (1):
- Private Practice of Dr. Andrew Blitzer, New York, New York, United States